CLINICAL TRIAL: NCT06168916
Title: AIMN Multicenter Study: 18 F-FDG PET-CT With or Without Contrast Medium in the Staging and Radiation of Lung Cancer?
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: POLMONE01
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET/CT with contrast medium in a single session. — Patients will undergo low dose PET/CT with FDG. Following the PET exam, a Standard CT with contrast medium will be acquired, using the CT tomography inserted inside the PET.

SUMMARY:
Accurate staging of patients with non-small cell cancer (NSCLC) is of fundamental importance both for the correct choice of treatment plan and for prognosis. Numerous studies have demonstrated the added value of co-registration of functional PET images and anatomical CT images using hybrid PET-CT tomographs and the consequent benefits on the choice of treatment in patients with NSCLC. Currently in most PET centers CT is performed with a "low dose" technique and is used exclusively as a transmissive source for attenuation correction and anatomical localization. The availability of new generation hybrid tomographs allows for "diagnostic" CT examinations (contrast CT) to be performed with a standard dose of radiation and with the use of intravenous and/or oral iodinated contrast medium (contrast medium). Little data is currently available on the added value of a PET-CT scan performed in a single session compared to PET-CT performed independently and, generally, subsequently to CT scan.

The objective of the study is to evaluate the ability to correctly define the accuracy in localizing and characterizing lung "lesions" in patients with confirmed NSCLC, in the staging or restaging phase, through the use of: PET-CT "low-dose" and PET contrast CT.

The effects of the two procedures on the patient's quality of life and on the costs incurred by the patient and the healthcare service will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically proven NSCLC, undergoing staging or restaging;
* plasma creatinine normal;

Exclusion Criteria:

* patients with lung microcytoma;
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with non-small cell lung cancer undergoing PET and contrast-enhanced CT during staging or restaging.
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2009-04-14 (Actual); Primary Completion 2010-11-11 (Actual); Study Completion 2010-11-11 (Actual)

PRIMARY OUTCOMES:
Use of PET and CT with contrast in a single session | 1 year
  In patients with confirmed NSCLC, evaluate the diagnostic accuracy of low dose PET-CT and contrast-enhanced PET CT

IPD SHARING:
Plan to Share IPD: No